CLINICAL TRIAL: NCT02689817
Title: Monitoring Physiologic Data in the Development of Pressure Ulcers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was withdrawn due to technical limitations to the device
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00093653
Record Dates: First submitted 2016-02-16; First posted 2016-02-24 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Pressure Ulcer; Signs and Symptoms
Keywords: Pressure ulcer; Monitoring; Pressure; Physiologic feedback
MeSH Terms: conditions — Pressure Ulcer; Signs and Symptoms | interventions — Transdermal Patch

STUDY DESIGN:
Masking Description: The investigator and outcomes assessors will be masked to the pressure data during the operating room and follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monitoring patch, no display (Experimental): Participants in this condition will receive a padded bandage that monitors pressure over time. In this arm, healthcare providers will not be able to view the pressure data collected.
  Interventions: Device: Patch

INTERVENTIONS:
Device: Patch — A bandage applied to the sacrum with pressure offloading characteristics and pressure monitoring components in a low-profile housing.

SUMMARY:
Hospital-acquired pressure ulcers (HAPUs) are a well-established serious complication of hospitalization that have serious consequences on patient morbidity and mortality as well as the cost of care. At the core of the problem for patient-centered targeted prevention of HAPUs is the lack of knowledge surrounding the magnitude and duration of pressure necessary to cause pressure ulcers, and the lack of immediate feedback on whether these interventions do anything to substantially offload at risk areas. Previous studies have been inconsistent in their findings of an association between duration of time and HAPU occurrence. While retrospectively this has been investigated, there is currently no substantial prospective, randomized study.

This study seeks to better understand the interface pressures between the patient and his or her support surface and how this relates to the development of pressure ulcers. The effect of patient characteristics and the relationship between total length of time on the operating table and pressure ulcer development will also be assessed.

The findings from this study will significantly add to strengthening the body of evidence regarding pressure ulcer development, specifically the relationship between the magnitude of interface pressure between the patient and the support surface for what duration of time leads to the development of a pressure ulcer. The results will provide critical insight into the physiologic targets healthcare providers should use to develop better pressure ulcer prevention programs, which could ultimately lead to a reduction in the incidence of pressure ulcers.

DETAILED DESCRIPTION:
Hospital-acquired pressure ulcers (HAPUs) are a well-established serious complication of hospitalization that have serious consequences on patient morbidity and mortality as well as the cost of care. Following CMS's changes to hospital reimbursements and penalization for hospitals with the highest rate of hospital-acquired complications, numerous quality improvement initiatives have been implemented. An overall reduction in the reported incidence of HAPUs from approximately 7 to 4.5% was observed, largely attributed to these interventions. Though there had been a drop in incidence, the overall number of hospitalized patients who develop HAPUs remains large and more recently HAPU frequency in hospitals has not continued to decrease, despite educational pressure ulcer prevention programs and clinical practice guidelines.

Due to the complications and costs associated with the development of a pressure ulcer, research has suggested that prevention is more effective than standard care. There are many current solutions for preventative interventions for HAPUs including leadership initiatives, data tracking, risk scales and many adjuvant pressure-offloading devices such as beds and mattress pads. Many of these devices have limited data supporting their effectiveness or are costly to implement in a purely prophylactic manner when current risk stratification methods fail to capture 60% of patients who go on to develop an ulcer. The vast majority of current preventative measures for pressure ulcers either seek to reduce the time a patient spends in one position or to reduce the magnitude of pressure that occurs on the high-risk areas for pressure ulcers. As such, manual repositioning (turning) is the most frequently used intervention as it is felt to be low-cost and part of standard care. Repositioning works by reducing or eliminating the interface pressure between the patient and the contact surface, but the standard recommendation on the 2 hour frequency were derived from animal studies and healthy volunteers. An expert consensus by Black et al. (2011) recommended the need for clinical decision-making based on the individual's needs and clinical situation when establishing a turning schedule, but there are very few objective tools that clinicians can use to make the decision.

At the core of the problem for patient-centered targeted prevention of HAPUs is the lack of knowledge surrounding the magnitude and duration of pressure necessary to cause pressure ulcers, and the lack of immediate feedback on whether these interventions do anything to substantially offload at risk areas. Previous studies have been inconsistent in their findings of an association between duration of surgery and HAPU occurrence, with results ranging from a negative association to a positive association.

This study seeks to better understand the interface pressures between the patient and his or her support surface and how this relates to the development of pressure ulcers. This data will provide critical insight into the physiologic targets healthcare providers should use to develop better pressure ulcer prevention programs and ultimately lead to a reduction in the incidence of pressure ulcers.

The primary outcome will be the interface pressure trend on the sacrum throughout the duration of time a patient is on the operating table and how that is correlated with pressure ulcer development. The effect of Braden scale score and other patient characteristics and the relationship between total length of time on the operating table and pressure ulcer development, and healthcare provider intervention in response to the pressure reading if in the second part of the study healthcare providers are not blinded to the pressure data.

This study will measure the interface pressure between a patient and his or her support surface in the operating room for prolonged (>2 hour) operative cases. Eligible patients will receive an adhesive padded bandage (similar to Mepilex Gentle Border) that collects interface pressure data. When the patient is being positioned in the operating room, this bandage will be applied to the sacrum. At the completion of the case the bandage will be removed and the status of the skin will be recorded and a photo of the sacrum will be taken for documentation. Skin status will be reassessed at 24 hours and at 1 week at regularly scheduled follow-ups with the surgeon. Pressure ulcer development will then be correlated with interface pressure characteristics during the operative case, using demographic data to check homogeneity between the experimental and control groups. If at interim analysis there is a clear relationship between a pressure threshold and pressure ulcer development, the second portion of the study will not blind healthcare providers to the live data. They would be able to see the pressure measurement and reposition the patient to effectively offload.

While retrospectively this has been investigated, there is currently no substantial prospective, randomized study. This study will significantly add to strengthening the body of evidence regarding pressure ulcer development, specifically the relationship between the magnitude of interface pressure between the patient and the support surface for what duration of time leads to the development of a pressure ulcer.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an operation that is scheduled to last more than 2 hours

Exclusion Criteria:

* Existing sacral pressure ulcer, undergoing a cardiac procedure, or inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Interface pressure (mmHg) over time (minutes) | Duration of the surgery (>120 min, <1440 min)
  The interface pressure trend on the sacrum throughout the duration of time a patient is on the operating table and how that is correlated with pressure ulcer development

SECONDARY OUTCOMES:
Pressure ulcer development | 1 week
  Skin will be checked immediately after the surgery and at 1 week using National Pressure Ulcer Advisory Panel (NPUAP) pressure ulcer staging system (grades I-IV).
Effect of Braden Scale | 1 week
  The relationship between interface pressure (mmHg), pressure ulcer development and Braden Scale Score (0-23).
Effect of Body Weight (kg) | 1 week
  The relationship between interface pressure (mmHg), pressure ulcer development and body weight (kilograms).
Effect of Body Mass Index (kg/m^2) | 1 week
  The relationship between interface pressure (mmHg), pressure ulcer development and body mass index (kg/m^2).
Effect of Age (years) | 1 week
  The relationship between interface pressure (mmHg), pressure ulcer development and age (years).
Effect of American Society of Anesthesiologists Score (I-IV) | 1 week
  The relationship between interface pressure (mmHg), pressure ulcer development and American Society of Anesthesiologists Score (I-VI).
Number of Repositioning events | Duration of the surgery (>2 h, <24 h)
  The number of times a patient is repositioned (defined by a greater than 50% change in the interface pressure (mmHg)) throughout the duration of the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Sacks, MD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berlowitz D, VanDeusen Lukas C, Parker V, Niederhauser A, Silver J, Logan C, Ayello E, Zulkowski K. 2012. Preventing Pressure Ulcers in Hospitals: A Toolkit for Improving Quality of Care. Rockville, MD: Agency for Healthcare Research and Quality; 2011. Rockville, MD: Agency for Healthcare Research and Quality.
- [Background] Black JM, Edsberg LE, Baharestani MM, Langemo D, Goldberg M, McNichol L, Cuddigan J; National Pressure Ulcer Advisory Panel. Pressure ulcers: avoidable or unavoidable? Results of the National Pressure Ulcer Advisory Panel Consensus Conference. Ostomy Wound Manage. 2011 Feb;57(2):24-37. PMID 21350270
- [Background] Feil M BJ. 2015. Hospital-Acquired Pressure Ulcers Remain a Top Patient Safety Concern for Hospitals in Pennsylvania. :1-10.
- [Background] Gillespie BM, Chaboyer WP, McInnes E, Kent B, Whitty JA, Thalib L. Repositioning for pressure ulcer prevention in adults. Cochrane Database Syst Rev. 2014 Apr 3;2014(4):CD009958. doi: 10.1002/14651858.CD009958.pub2. PMID 24700291
- [Background] Hommel A, Bjorkelund KB, Thorngren KG, Ulander K. Nutritional status among patients with hip fracture in relation to pressure ulcers. Clin Nutr. 2007 Oct;26(5):589-96. doi: 10.1016/j.clnu.2007.06.003. Epub 2007 Jul 26. PMID 17662510
- [Background] Houwing R, Rozendaal M, Wouters-Wesseling W, Buskens E, Keller P, Haalboom J. Pressure ulcer risk in hip fracture patients. Acta Orthop Scand. 2004 Aug;75(4):390-3. doi: 10.1080/00016470410001132-1. PMID 15370580
- [Background] KOSIAK M. Etiology and pathology of ischemic ulcers. Arch Phys Med Rehabil. 1959 Feb;40(2):62-9. No abstract available. PMID 13618101
- [Background] KOSIAK M. Etiology of decubitus ulcers. Arch Phys Med Rehabil. 1961 Jan;42:19-29. No abstract available. PMID 13753341
- [Background] Lindholm C, Sterner E, Romanelli M, Pina E, Torra y Bou J, Hietanen H, Iivanainen A, Gunningberg L, Hommel A, Klang B, Dealey C. Hip fracture and pressure ulcers - the Pan-European Pressure Ulcer Study - intrinsic and extrinsic risk factors. Int Wound J. 2008 Jun;5(2):315-28. doi: 10.1111/j.1742-481X.2008.00452.x. PMID 18494637
- [Background] McInnes E, Jammali-Blasi A, Bell-Syer SE, Dumville JC, Middleton V, Cullum N. Support surfaces for pressure ulcer prevention. Cochrane Database Syst Rev. 2015 Sep 3;2015(9):CD001735. doi: 10.1002/14651858.CD001735.pub5. PMID 26333288
- [Background] Meddings J. Using administrative discharge diagnoses to track hospital-acquired pressure ulcer incidence--limitations, links, and leaps. Jt Comm J Qual Patient Saf. 2015 Jun;41(6):243-5. doi: 10.1016/s1553-7250(15)41033-5. No abstract available. PMID 25990889
- [Background] Padula WV, Makic MB, Mishra MK, Campbell JD, Nair KV, Wald HL, Valuck RJ. Comparative effectiveness of quality improvement interventions for pressure ulcer prevention in academic medical centers in the United States. Jt Comm J Qual Patient Saf. 2015 Jun;41(6):246-56. doi: 10.1016/s1553-7250(15)41034-7. PMID 25990890
- [Background] Padula WV, Makic MB, Wald HL, Campbell JD, Nair KV, Mishra MK, Valuck RJ. Hospital-Acquired Pressure Ulcers at Academic Medical Centers in the United States, 2008-2012: Tracking Changes Since the CMS Nonpayment Policy. Jt Comm J Qual Patient Saf. 2015 Jun;41(6):257-63. doi: 10.1016/s1553-7250(15)41035-9. PMID 25990891
- [Background] Peich S, Calderon-Margalit R. Reduction of nosocomial pressure ulcers in patients with hip fractures: a quality improvement program. Int J Health Care Qual Assur Inc Leadersh Health Serv. 2004;17(2-3):75-80. doi: 10.1108/09526860410526682. PMID 15301263
- [Background] Qaseem A, Mir TP, Starkey M, Denberg TD; Clinical Guidelines Committee of the American College of Physicians. Risk assessment and prevention of pressure ulcers: a clinical practice guideline from the American College of Physicians. Ann Intern Med. 2015 Mar 3;162(5):359-69. doi: 10.7326/M14-1567. PMID 25732278
- [Background] Ratliff CR; WOCN. WOCN's evidence-based pressure ulcer guideline. Adv Skin Wound Care. 2005 May;18(4):204-8. doi: 10.1097/00129334-200505000-00009. No abstract available. PMID 15920372
- [Background] Reddy M, Gill SS, Rochon PA. Preventing pressure ulcers: a systematic review. JAMA. 2006 Aug 23;296(8):974-84. doi: 10.1001/jama.296.8.974. PMID 16926357
- [Background] VanGilder C, Amlung S, Harrison P, Meyer S. Results of the 2008-2009 International Pressure Ulcer Prevalence Survey and a 3-year, acute care, unit-specific analysis. Ostomy Wound Manage. 2009 Nov 1;55(11):39-45. PMID 19934462